CLINICAL TRIAL: NCT07013929
Title: Spyral InSight Early Clinical Feasibility Study
Brief Title: Spyral InSight Study
Acronym: Spyral InSight
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT24037
Record Dates: First submitted 2025-04-18; First posted 2025-06-10 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Vascular Diseases; Cardiovascular Diseases
Keywords: Hypertension; Cardiovascular Diseases; Vascular Diseases; Denervation; Renal Denervation
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Renal nerve stimulation performed prior to and post renal artery denervation (RDN) (Experimental)
  Interventions: Device: Renal nerve stimulation

INTERVENTIONS:
Device: Renal nerve stimulation — Renal nerve stimulation will be performed prior to and post renal denervation.

SUMMARY:
The purpose of the Spyral InSight Early Clinical Feasibility Study is to characterize the physiological response to renal nerve stimulation (RNS) in humans prior to and post renal denervation.

DETAILED DESCRIPTION:
This study is exploratory in nature and an early-stage clinical assessment that will evaluate procedural and long-term safety of renal nerve stimulation (RNS) when performed prior to and post renal artery denervation (RDN) with the Symplicity Spyral system, with follow-up at 1, 3, 6 and 12 months.

There is no pre-specified primary endpoint. However, the objectives of the Spyral InSight ECF study are as follows:

* To assess safety of RNS when performed prior to and post RDN.
* To characterize and quantify the physiological response to renal nerve stimulation in humans undergoing renal denervation per approved labeling.

ELIGIBILITY:
Inclusion Criteria:

1. 20 - 70 years of age
2. Office SBP ≥150 mmHg and <180 mmHg and DBP ≥90 mmHg
3. Individual is prescribed with one, two, or three antihypertensive medication classes
4. 24-hour ABPM average of SBP ≥135 and <170 mmHg at Baseline

Exclusion Criteria:

1. Prior renal denervation.
2. Individual lacks appropriate renal artery Anatomy
3. Has a renal artery stent
4. Individual has an estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73m2
5. Individual is taking SGLT2 inhibitors or GLP-1 agonists
6. Individual requires chronic oxygen support or mechanical ventilation
7. Primary pulmonary hypertension.
8. Secondary cause of hypertension
9. Pregnant, nursing or planning to become pregnant during the study.
10. Individual has a documented condition that would prohibit or interfere with ability to obtain an accurate blood pressure measurement
11. Individual is currently taking anti-mineralocorticoid drugs.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Through study completion, from enrollment to 12-month follow-up
End-stage renal disease | Through study completion, from enrollment to 12-month follow-up
Myocardial infarction | Through study completion, from enrollment to 12-month follow-up
Incidence of stroke | Through study completion, from enrollment to 12-month follow-up
Hospitalization for hypertensive crisis not related to non-adherence with medications | Through study completion, from enrollment to 12-month follow-up
Significant embolic event resulting in end-organ damage | Through study completion, from enrollment to 12-month follow-up
Renal artery intervention | Through study completion, from enrollment to 12-month follow-up
New renal artery stenosis >70%, confirmed by angiography and as determined by the angiographic core lab | Through study completion, from enrollment to 12-month follow-up
Vascular complications | Through study completion, from enrollment to 12-month follow-up
Major bleeding according to TIMI definition | Through study completion, from enrollment to 12-month follow-up
Prolonged renal vasoconstriction requiring intervention | Through study completion, from enrollment to 12-month follow-up
Contrast induced nephropathy | Through study completion, from enrollment to 12-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.